CLINICAL TRIAL: NCT00833937
Title: A Relative Bioavailability Study of Zolpidem Tartrate 10 mg Tablets Under Non-Fasting Conditions
Brief Title: Zolpidem Tartrate 10 mg Tablets Under Non-Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: B016540
Record Dates: First submitted 2009-01-30; First posted 2009-02-02 (Estimated); Results first posted 2009-08-18 (Estimated); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Zolpidem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zolpidem (Experimental): Zolpidem Tartrate 10 mg Tablet (test) dosed in first period followed by Ambien® 10 mg Tablet (reference) dosed in second period
  Interventions: Drug: Zolpidem 10 mg tablets
- Ambien® (Active Comparator): Ambien® 10 mg Tablet (reference) dosed in first period followed by Zolpidem Tartrate 10 mg Tablet (test) dosed in second period
  Interventions: Drug: AMBIEN® 10 mg tablets

INTERVENTIONS:
Drug: Zolpidem 10 mg tablets — 1 x 10 mg
  Arms: Zolpidem
Drug: AMBIEN® 10 mg tablets — 1 x 10 mg
  Arms: Ambien®

SUMMARY:
The objective of this study is to compare the relative bioavailability of Zolpidem tartrate 10 mg tablets (manufactured by TEVA Pharmaceutical Industries, Ltd. and distributed by TEVA Pharmaceuticals USA) with that of AMBIEN® tablets(G.D. Searle & Co.) in healthy, adult, non-smoking subjects under non-fasting conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* All subjects selected for this study will be non-smokers at least 18 years of age. Subjects will have a BMI (body mass index) of 30 or less.

Exclusion Criteria:

* Subjects with a significant recent history of chronic alcohol consumption, drug addiction, or serious gastrointestinal, renal, hepatic or cardiovascular disease, tuberculosis, epilepsy, asthma, diabetes, psychosis or glaucoma will not be eligible for this study.
* Subjects whose clinical laboratory test values are greater than 20% outside the normal range may be retested. If the clinical values are outside the range on retesting, the subject will not be eligible to participate in the study unless the clinical investigator deems the result to not be significant.
* Subjects who have a history of allergic responses to the class of drug being tested will be excluded from the study.
* Subjects who use tobacco in any form will not be eligible to participate in the study. Three months abstinence is required.
* All subjects will have urine samples assayed for the presence of drugs of abuse as part of the clinical laboratory screening procedures and at each dosing period check-in. Subjects found to have urine concentrations of any of the tested drugs will not be allowed to participate.
* Subjects should not have donated blood and/or plasma for at least thirty (30) days prior to the first dosing of the study.
* Subjects who have taken any investigational drug within thirty (30) days prior to the first dosing of the study will not be allowed to participate.
* Female subjects who are pregnant, breast-feeding, or who are likely to become pregnant during the study will not be allowed to participate. Female subjects of child bearing potential must either abstain from sexual intercourse or use a reliable barrier method (e.g. condom, IUD) of contraception during the course of the study (first dosing until last blood collection) or they will not be allowed to participate. Subjects who have used implanted or injected hormonal contraceptives anytime during the 180 days prior to study dosing or oral hormonal contraceptives with in 14 days of dosing will not be allowed to participate.
* All Female subjects will be screened for pregnancy at check-in each study period. Subjects with positive or inconclusive results will be withdrawn from the study.
* Subjects who do not tolerate venipuncture will not be allowed to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2002-03; Primary Completion 2002-03 (Actual); Study Completion 2002-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Ann Kennedy, M.D., Principal Investigator — Novum Pharmaceuticals Research Services
Locations (2):
- United States (2):
  - Novum Pharmaceutical Research Services, Pittsburgh, Pennsylvania
  - Bioassay Laboratory, Inc., Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Zolpidem (Test) First: Zolpidem Tartrate 10 mg Tablet (test) dosed in first period followed by Ambien® 10 mg Tablet (reference) dosed in second period
- Ambien® (Reference) First: Ambien® 10 mg Tablet (reference) dosed in first period followed by Zolpidem Tartrate 10 mg Tablet (test) dosed in second period
Period: First Intervention
Arm/Group | Zolpidem (Test) First | Ambien® (Reference) First
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Washout
Arm/Group | Zolpidem (Test) First | Ambien® (Reference) First
Started | 12 | 12
Completed | 11 | 12
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Second Intervention
Arm/Group | Zolpidem (Test) First | Ambien® (Reference) First
Started | 11 | 12
Completed | 11 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zolpidem (Test) First | Ambien® (Reference) First | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 11 | 10 | 21
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 9 | 7 | 16
  Black | 2 | 4 | 6
  Hispanic | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Concentration
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 24 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Zolpidem: Zolpidem Tartrate 10 mg Tablet (test) dosed in either period
- Ambien®: Ambien® 10 mg Tablet (reference) dosed in either period
Arm/Group | Zolpidem | Ambien®
Number analyzed (Participants) | 23 | 23
ng/mL | 117.313 (42.878) | 116.452 (40.419)
Statistical Analysis 1: Comparison: Zolpidem vs Ambien®; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Ratio of Geometric Means = 99.7, 90% CI [93.9 to 106] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

2. Primary Outcome: AUC0-inf - Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated)
Description: Bioequivalence based on AUC0-inf
Time Frame: Blood samples collected over 24 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Zolpidem | Ambien®
Number analyzed (Participants) | 23 | 23
ng*h/mL | 541.580 (279.254) | 543.732 (273.918)
Statistical Analysis 1: Comparison: Zolpidem vs Ambien®; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Ratio of Geometric Means = 97.8, 90% CI [92.6 to 103] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

3. Primary Outcome: AUC0-t - Area Under the Concentration-time Curve From Time Zero to Time of Last Non-zero Concentration (Per Participant)
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 24 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Zolpidem | Ambien®
Number analyzed (Participants) | 23 | 23
ng*h/mL | 530.272 (271.461) | 531.866 (265.350)
Statistical Analysis 1: Comparison: Zolpidem vs Ambien®; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Ratio of Geometric Means = 97.9, 90% CI [92.7 to 103] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator is not permitted to discuss or publish trial results.